CLINICAL TRIAL: NCT07330284
Title: Adjunctive Cold Water Irrigation Added to Rectal Indomethacin for Prevention of Post- Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Brief Title: Cold Water Irrigation Therapy as an Adjunct to Indomethacin for Post-Endoscopic Retrograde Cholangiopancreatography(ERCP) Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Reza Hejazi, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KU-IIS-RH-2025-01
Record Dates: First submitted 2025-11-06; First posted 2026-01-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pancreatitis; ERCP Surgery
Keywords: Cold Water; Prevention; ERCP; Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Water (Experimental): • Cold Water Irrigation of the Papilla: Participants randomized to the experimental arm will receive 250 mL of refrigerated water (target temperature 4-8 °C) in five 50 mL aliquots directed toward the papilla, with duodenal aspiration after each aliquot.
  Interventions: Procedure: Cold water
- Warm water (Placebo Comparator): • Control Intervention: Participants randomized to the control group will receive 250 mL of room-temperature water in identical increments and delivery.
  Interventions: Procedure: Warm water

INTERVENTIONS:
Procedure: Cold water — Rectal indomethacin plus cold water irrigation
  Arms: Cold Water
Procedure: Warm water — Rectal indomethacin plus room-temperature water irrigation
  Arms: Warm water

SUMMARY:
This study is designed to learn whether rinsing the papilla with cold water at the end of an ERCP procedure, in addition to standard medicine, can help lower the chance of developing pancreatitis, which is the most common major complication after ERCP.

DETAILED DESCRIPTION:
Study design:

This is an investigator-initiated, single-center, triple-blind, parallel-group, randomized controlled superiority trial. Participants will be randomized 1:1 to receive either (1) rectal indomethacin plus cold water irrigation or (2) rectal indomethacin plus room-temperature water irrigation. The study is designed to evaluate whether cold water irrigation provides additive benefit in reducing the incidence of post-ERCP pancreatitis (PEP) compared with standard therapy.

Eligible patients (≥20 years, native papilla) undergoing ERCP at University of Kansas Medical Center (KUMC) will be identified during pre-procedure evaluation. Written informed consent will be obtained prior to the procedure.

Baseline Data Collection: Demographic data, relevant medical history, ERCP indication, and risk factors for PEP will be recorded before the procedure.

All patients receive a 100 mg rectal indomethacin suppository at the completion of ERCP.

Participants are randomized to receive either 250 mL of cold water (experimental arm) or room-temperature water (control arm) directed toward the papilla in five 50 mL aliquots, with aspiration between each injection.

Monitoring During ERCP: Continuous monitoring of heart rate, non-invasive blood pressure, oxygen saturation, and sedation status will be performed throughout the procedure per standard of care.

Post-Procedure Monitoring: Patients will be monitored in the recovery unit and inpatient setting as clinically indicated. Laboratory tests (amylase, lipase, Complete Blood Count (CBC), metabolic panel) will be obtained if patients develop post-procedure abdominal pain or clinical suspicion of pancreatitis.

Risk Minimization, Drugs/Devices, and Source Records :

• Risk Minimization: All patients receive guideline-recommended NSAID prophylaxis (indomethacin).Cold water irrigation volume and temperature are standardized to avoid mucosal injury or systemic effects. Experienced endoscopists will perform all procedures. Patients will be closely monitored during and after ERCP for early recognition of adverse events.

• Drugs/Devices: Rectal indomethacin (100 mg suppository) - FDA-approved NSAID, used off-label for PEP prevention.

Sterile water for irrigation (cold or room temperature) - procedural adjunct, not investigational.

• Source Records: Electronic medical record (Epic) for demographics, labs, and hospital course. Procedure reports and nursing documentation. Case report forms (CRFs) and study data collection sheets maintained in a secure REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* Native papilla present.
* Undergoing ERCP for diagnostic or therapeutic indications.
* Able to provide informed consent.

Exclusion Criteria:

* Post-operative reconstructed intestinal tract other than Billroth I reconstruction.
* Acute pancreatitis at the time of ERCP.
* Chronic pancreatitis.
* Pancreatic head cancer with occlusion of the main pancreatic duct.
* Existing pancreatic duct stent or need for prophylactic pancreatic duct stenting during the index ERCP.
* Known contraindications or allergy to indomethacin or other NSAIDs.
* Significant renal impairment (eGFR < 30 mL/min/1.73m²).
* Active peptic ulcer disease or history of NSAID-induced gastrointestinal bleeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-ERCP Pancreatitis (PEP) between the cold water and control groups | approximately 24-36 months.
  The incidence of post-ERCP pancreatitis (PEP) is defined according to established consensus criteria as new or worsened abdominal pain persisting for at least 24 hours after ERCP, accompanied by serum amylase or lipase levels ≥3 times the upper limit of normal at approximately 24 hours post-procedure, and necessitating hospital admission or prolongation of planned observation.

SECONDARY OUTCOMES:
Severity of post-ERCP pancreatitis | Up to 7 days post-ERCP
  Severity of post-ERCP pancreatitis will be classified per the Revised Atlanta Classification (mild, moderate, or severe), based on organ failure, its duration, and local or systemic complications, with follow-up through 7 days post-ERCP

OTHER OUTCOMES:
Length of Hospital Stay Following ERCP | Up to 7 days post-ERCP
  Total number of days hospitalized from the day of ERCP through Day 7 post-ERCP.
Requirement for Additional Interventions Related to Post-ERCP Pancreatitis | Up to 7 days post-ERCP
  Proportion of participants requiring additional interventions related to post-ERCP pancreatitis, including intensive care unit (ICU) admission or surgical or radiologic intervention.
Incidence of Other ERCP-Related Adverse Events | Up to 7 days post-ERCP
  Proportion of participants experiencing ERCP-related adverse events other than post-ERCP pancreatitis, including bleeding, perforation, cholangitis, or cardiopulmonary complications.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Hejazi, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
All personnel involved in this project are the University of Kansas (KU)-affiliated physicians/researchers; therefore, there are no anticipated issues regarding the sharing of individual participant data (IPD).